CLINICAL TRIAL: NCT04893070
Title: Impact of SARS-CoV-2 (COVID-19) Infection, Treated in Ambulatory Care, on Long-term Quality of Life in a Parisian Military Population
Acronym: COVIDAMBUCMA1
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-COVID19-38; 2021-A01038-33 (Other: IDRCB)
Record Dates: First submitted 2021-05-11; First posted 2021-05-19 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: SARS-CoV2 Infection; Covid19
Keywords: Quality of life
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID+: Questionnaires on COVID-19 symptomatology and quality of life
  Interventions: Other: Questionnaires COVID+
- COVID-: Questionnaires on quality of life
  Interventions: Other: Questionnaires COVID-

INTERVENTIONS:
Other: Questionnaires COVID+ — * 1 questionnaire on COVID-19 symptomatology and quality of life 12 months after COVID-19 first symptoms
  * 1 questionnaire on quality of life 18 months after COVID-19 first symptoms
  Groups: COVID+
Other: Questionnaires COVID- — * 1 questionnaire on quality of life at enrollment
  * 1 questionnaire on quality of life 6 months after enrollment
  Groups: COVID-

SUMMARY:
In April 2020, a meta-analysis on the long-term sequelae of respiratory syndromes related to seasonal coronaviruses (SARS and MERS) showed a significant alteration in quality of life, with in particular a decrease in physical and emotional capacities and a deterioration of social life. An improvement of the quality of life is evidenced after 6 months but without reaching the level usually observed in healthy people. The impact of SARS-CoV-2 infection on quality of life can be explained by the persistence of pleomorphic symptoms in the medium to long term. In the military population, the majority of SARS-CoV-2 cases present minor to moderate forms of the disease. Military personnel have living conditions that differ from those of the general population, in particular because of their geographic mobility, which may be responsible for isolation from the family. This isolation can be regular (we speak of "geographical celibacy" when the soldier is posted in a geographical area far from the family unit) and/or occasional, during missions on the national territory or outside. This singularity justifies a study on the impact of SARS-CoV-2 (COVID-19) infection on the quality of life in this specific population.

ELIGIBILITY:
Inclusion Criteria:

* Military personnel
* COVID+: diagnosed with COVID-19 and managed in ambulatory care since March 14th, 2020
* COVID-: not having been infected with SARS-CoV-2

Exclusion Criteria:

* Hospitalized for COVID-19
* Having received a treatment against COVID-19 (other than paracetamol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is composed of military staff followed at the 1st Centre Médical des Armées (Paris, France) who have suffered from COVID-19 and were managed in ambulatory care (COVID+ group) and who have not been infected by SARS-CoV-2 (COVID- group).
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Long-term quality of life (mental component) | 18 months after COVID-19 first symptoms
  Mental Component Score (MCS) of the SF-36 questionnaire. The MCS ranges from 0 (bad quality of life) to 100 (good quality of life).

SECONDARY OUTCOMES:
Long-term quality of life (physical component) | 18 months after COVID-19 first symptoms
  Physical Component Score (PCS) of the SF-36 questionnaire. The PCS ranges from 0 (bad quality of life) to 100 (good quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- 1er Centre Médical des Armées, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided